CLINICAL TRIAL: NCT04719559
Title: Combined Use of Fractional Laser and Steroid Ointment to Improve the Old Scar After Thyroidectomy
Brief Title: Fractional Laser and Steroid Ointment to Improve the Old Scar After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201800241A3
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Thyroid; Wound; Steroid Acne
MeSH Terms: conditions — Thyroid Diseases; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Thyroidectomy Hypertrophic Scar (Other): Patients had all presented a persistent hypertrophic scar at the neck region for more than 1 year after their thyroidectomy.
  Interventions: Device: Laser-assisted drug delivery

INTERVENTIONS:
Device: Laser-assisted drug delivery — All patients received treatment using the same protocol with the same fractional ablative carbon dioxide laser (eCO2 PlusTM, manufactured by Lutronic, South Korea). Each patient was applied with Lidopin 5% cream (Panion & BF Biotech Inc.), which remained on the scar for 30 min for pain relief before each laser course. Later, the Lidopin 5% cream was gently removed using a normal saline-rinsed gauze, and the scar was treated with a fractional ablative carbon dioxide laser with two passes under a 10,600 nm wavelength, 120 mm spot size, pulse energy of 50 mJ, 30 W of power, and a density of 200. A topical steroid cream (clobetasol propionate, 0.05%) was evenly applied on the scar gently back and forth using a cotton swab immediately after the laser treatment. The patients underwent five full courses by the same doctor according to the same protocol, with each course given 4 weeks apart.

SUMMARY:
This clinical study was conducted to assess the effects of LADD combined with a fractional ablative carbon dioxide laser and a topical steroid for the treatment of post-thyroidectomy hypertrophic scars.

DETAILED DESCRIPTION:
Thyroidectomy results in unsightly scarring at the anterior neck of the patient. A clinical study was conducted to assess the effectiveness of five courses, applied every 4 weeks, of laser-assisted drug delivery (LADD) combining a fractional ablative carbon dioxide laser and topical 0.05% clobetasol propionate to the treatment of post-thyroidectomy hypertrophic scars in patients. Assessments of the scars by the patient themselves according to the patient and observer scar assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients had presented a persistent hypertrophic scar at the neck region for more than 1 year after their thyroidectomy.

Exclusion Criteria:

* Systemic chronic disease or a history of autoimmune disease or human immunodeficiency virus infections.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Self-assessment by patients before treatment | before first treatment
  For each patient's self-assessment before the first treatment, we adopted the patient and observer scar assessment scale (POSAS)18, with a range of 1-10 for representing the severity of the itchiness, pain, color, softness, thickness, irregularity, and distorted appearance of the scar.
Self-assessment by patients after treatment | 1 year after the first treatment
  For each patient's self-assessment1 year after the first treatment, we adopted the patient and observer scar assessment scale (POSAS)18, with a range of 1-10 for representing the severity of the itchiness, pain, color, softness, thickness, irregularity, and distorted appearance of the scar.
Doctor evaluations using the POSAS scoring range of 1-10 | 1 year after the first treatment
  Four doctors participated as observers of the clinical outcomes. One of the doctors carried out all treatments and evaluated seven parameters, namely, vascularity, pigmentation, thickness, relief, pliability, surface area, and overall opinion based on the POSAS using a scoring range of 1-10, from normal to worst conditions 1 year after the first treatment. The remaining three doctors acted as observers to evaluate the general appearances of the scars based on photographs captured by the same photographer with the same camera 1 year after the first treatment. They then rated the scar on a score of 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan